CLINICAL TRIAL: NCT00520949
Title: Quadruple Therapy Using Esomeprazole, Colloidal Bismuth Subcitrate, Amoxicillin-Clavulanate, and Furazolidone in Patients Who Failed to Eradicate H. Pylori With Triple Therapy
Brief Title: Quadruple Therapy for Triple Therapy Resistant Helicobacter Pylori Infection
Acronym: QT-Hp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Dr Zaigham Abbas, The Aga Khan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 609-Med
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Treatment of Helicobacter Pylori
Keywords: H.pylori; Triple therapy failure; Quadruple therapy
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Furazolidone; bismuth tripotassium dicitrate; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quadruple Therapy (Experimental)
  Interventions: Drug: Augmentin (Amoxicillin-clavulanic); Drug: Furoxone (furazolidone); Drug: Cebes (colloidal bismuth subcitrate); Drug: Esso (esomeprazole)

INTERVENTIONS:
Drug: Augmentin (Amoxicillin-clavulanic) — Amoxicillin-clavulanic acid 1 gram b.i.d
Drug: Furoxone (furazolidone) — furazolidone 200 mg b.i.d
Drug: Cebes (colloidal bismuth subcitrate) — colloidal bismuth subcitrate 240 mg b.i.d
Drug: Esso (esomeprazole) — esomeprazole 40 mg b.i.d for 14 days

SUMMARY:
Triple therapy, a combination of proton pump inhibitor with two antibiotics, is the gold standard for anti-Helicobacter pylori treatment. Usual antibiotics are clarithromycin, and either amoxicillin or one of the nitroimidazoles (metronidazole). However, there is an increasing evidence of H. pylori resistance to classical triple therapy. Another reason for this failure being low patient compliance with treatment. A regimen useful in one geographical area may not be effective or practical in another area. The aim of this study was to eradicate H. pylori infection resistant to triple therapy, establish the efficacy and safety of a 14-day therapeutic regimen to eradicate of H. pylori in patients who have failed with the classical triple therapy (omeprazole, clarithromycin and amoxicillin) given for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given by the patient
* Patients known to have H. pylori infection diagnosed by histopathology, rapid urease test and urea breath test
* Failure to respond to classical triple regime of amoxicillin 1gram, clarithromycin 500mg and omeprazole 20mg twice a day for 10-14 days as documented by repeat urea breath test done one month after eradication therapy

Exclusion Criteria:

* Evidence of any malignancy, gastric outlet syndrome, history of gastric surgery, chronic liver disease, severe chronic renal failure, or any major co-morbidity.
* known or suspected hypersensitivity to the medication used in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Eradication of H. pylori infection resistant to triple therapy. | 6 weeks

SECONDARY OUTCOMES:
Safety of the quadruple therapy | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zaigham Abbas, FACG, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Abbas Z, Yakoob J, Abid S, Jafri W, Islam M, Azam Z, Hilal I. Furazolidone, co-amoxiclav, colloidal bismuth subcitrate, and esomeprazole for patients who failed to eradicate Helicobacter pylori with triple therapy. Dig Dis Sci. 2009 Sep;54(9):1953-7. doi: 10.1007/s10620-008-0582-6. Epub 2008 Dec 5. PMID 19058002